CLINICAL TRIAL: NCT00002889
Title: PROGNOSTIC SIGNIFICANCE OF ENDORECTAL MRI IN PREDICTING OUTCOME AFTER COMBINED RADIATION AND ANDROGEN SUPPRESSION FOR PROSTATE CANCER: A PROSPECTIVE PHASE II STUDY
Brief Title: Radiation Therapy With Androgen Suppression in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9682; U10CA031946 (NIH); CLB-9682; CDR0000065212 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: flutamide
Drug: goserelin
Drug: leuprolide acetate
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Imaging procedures such as MRI may improve the ability to determine the response of prostate tumors to therapy.

PURPOSE: Phase II trial to study MRI results in patients with prostate cancer that has been treated with radiation therapy plus androgen suppression therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Establish whether changes between baseline and 2-month post androgen suppression endorectal coil MRI results predict for biochemical control following radiotherapy with androgen suppression in patients with adenocarcinoma of the prostate.

OUTLINE: Patients undergo a baseline endorectal coil MRI, followed by total androgen suppression (TAS) with either leuprolide IM or subcutaneous goserelin once a month plus oral flutamide 3 times a day for 2 months. Patients then receive a second endorectal coil MRI, followed by 2 months of external-beam radiotherapy plus TAS. Patients may receive an additional 2 months of TAS at the discretion of the treating physician. Patients are followed every 6 months for 3 years, then yearly thereafter.

PROJECTED ACCRUAL: Approximately 180 patients (approximately 60 per year) will be accrued for this study over a 34 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate AJCC stage T1b-T4b, N0 or Nx, M0 Transrectal, transperineal, or transurethral biopsy required

PATIENT CHARACTERISTICS: Age: 30 and over Performance status: CALGB 0-2 Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: The following may increase the risk of protocol treatment: Serious intercurrent medical illness that might compromise patient safety Active acute infection requiring antibiotics Suppression therapy for chronic urinary tract infection allowed Uncontrolled or severe cardiovascular disease Psychiatric conditions that prevent compliance or informed consent

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for carcinoma of the prostate Endocrine therapy: No prior androgen deprivation therapy (medical or surgical) Radiotherapy: No prior radiation therapy for carcinoma of the prostate Surgery: No prior surgical androgen deprivation therapy

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 1997-05; Primary Completion 2004-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2 years post tx

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V. D'Amico, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Joint Center for Radiation Therapy, Boston, Massachusetts
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Result] D'Amico AV, Halabi S, Tempany C, Titelbaum D, Philips GK, Loffredo M, McMahon E, Sanford B, Vogelzang NJ, Small EJ; Cancer and Leukemia Group B. Tumor volume changes on 1.5 tesla endorectal MRI during neoadjuvant androgen suppression therapy for higher-risk prostate cancer and recurrence in men treated using radiation therapy results of the phase II CALGB 9682 study. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):9-15. doi: 10.1016/j.ijrobp.2007.09.033. Epub 2007 Nov 26. PMID 18037582
- [Result] D'Amico AV, Halabi S, Vollmer R, Loffredo M, McMahon E, Sanford B, Archer L, Vogelzang NJ, Small EJ, Kantoff PW; Cancer and Leukemia Group B. p53 protein expression status and recurrence in men treated with radiation and androgen suppression therapy for higher-risk prostate cancer: a prospective phase II Cancer and Leukemia Group B Study (CALGB 9682). Urology. 2008 May;71(5):933-7. doi: 10.1016/j.urology.2007.11.005. Epub 2008 Feb 21. PMID 18291508
- [Result] D'Amico AV, Halabi S, Tempany C, et al.: Changes on endorectal MRI during neoadjuvant hormonal therapy for prostate cancer and biochemical outcome in men managed using radiation therapy: a prospective phase II Cancer and Leukemia Group B study. [Abstract] J Clin Oncol 25 (Suppl 18): A-5072, 252s, 2007.